CLINICAL TRIAL: NCT00608452
Title: A Prospective Study of The Prevalence and Significance of Paraneoplastic Autoantibodies in Small Cell Lung Cancer and Cancer of The Breast, Ovary, Hodgkin's Disease, Neuroblastoma and Other Cancers
Brief Title: Prevalence+Significance of Paraneoplastic Autoantibodies in Many Cancers
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Posner, Jerome, M /Principal Investigator, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 95-046
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Lung Cancer; Ovarian Cancer; Breast Cancer; Hodgkin's Disease; Neuroblastoma
Keywords: Lung; Ovarian; Breast; Hodgkin's
MeSH Terms: conditions — Lung Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Hodgkin Disease; Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for autoantibody determinations and HLA typing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Symptom Assessment Scale

INTERVENTIONS:
Other: Symptom Assessment Scale — * Memorial Symptom Assessment Scale
  * History and neurologic examination

SUMMARY:
You may have a type of cancer associated with "antineuronal antibodies" in your blood.

Antibodies are substances made by the immune system. They are used by the body to fight infections and other diseases. Antineuronal antibodies are antibodies that react with nerve cells but they also react with some tumors. We believe that the immune system makes these antibodies to fight the cancer. In some patients with these antibodies, the tumor is smaller than in patients who have no antibodies. Sometimes, with a very strong antibody test, patients may develop neurologic problems such as weakness, numbness or memory loss. One purpose of this study is to determine if a patient with cancer and a positive antineuronal antibody blood test has a smaller tumor and responds better to treatment than a patient with cancer and a negative test. Another purpose of this study is to determine whether patients with a positive antibody test develop neurologic problems such as weakness, numbness or memory loss.

We will measure your blood for several different kinds of antibodies in addition to antineuronal antibodies to determine if the presence of antibodies predicts "prognosis", i.e. smaller tumor and better response to treatment, or predicts the development of neurologic problems.

No tissue samples are required for this study. However, if tissue or sputum is obtained by your oncologist for diagnostic purposes, we will ask your doctors or the pathology department to provide us with samples of these specimens. This will not involve any additional surgery or discomfort to you.

DETAILED DESCRIPTION:
Objectives:

To determine prospectively the prevalence and specificity of anti-Hu and other paraneoplastic antibodies in patients with small cell lung cancer (SCLC) and other cancers including, but not limited to, ovarian cancer, breast cancer and Hodgkin's disease / the prevalence of other autoimmune antibodies in patients with SCLC and other cancers including but not limited to anti-nuclear antibodies, anti-P53 antibodies, rheumatoid factor and anti-calcium channel antibodies /the prevalence and significance of antibodies against a LEMS-related antigen (MysB)/whether the production of autoantibodies including anti-Hu antibodies is related to patient MHC phenotype.

* To examine tumor specimens and other available tissues (sputum and bone marrow, if possible) for the presence of Hu antigen-expressing cells, and/or cells expressing other paraneoplastic antigens/patients with SCLC and other cancers for the development of neurologic signs, paraneoplastic or otherwise.
* Attempts will be made to evaluate all patients at the time of initial consultation by the primary oncologist. If this is not possible, attempts will be made to obtain the neurological evaluation at the time of the next visit with the oncologist, or in case of inpatients, during the patient's admission. A complete history and neurologic examination will be performed at that time by the neurologist with documentation of signs and symptoms. The patient will be given the Memorial Symptom Assessment Scale to complete (see attached).
* At initial evaluation, blood will be obtained for the following laboratory studies including but not limited to (for children the amount of blood drawn will be no more than 5 cc per Kg for each visit): A) Rheumatoid Factor and Anti-nuclear, anti-thyroglobulin, anti-microsomal, anti-Ro, and antip53 antibodies. B) HLA Typing (HLA-ABC, IEF, Class II DNA) and lymphocyte analysis C) Anti-neuronal antibodies, including HuD, HuC and HeI-N1, anti-Yo, anti-Ri, anti-Tr antibodies D) LEMS-associated antibodies (MysB antibodies)
* At follow-up (approximately every 4 months) appointments, blood samples will be obtained for the following studies, including but not limited to, anti-neuronal antibodies HuC and HeI-N1) and LEMS-associated antibodies (MysB antibodies).
* Tissue samples obtained at diagnosis or during the course of treatment (tumor resection or biopsy, sputum collections or bone marrow aspirations) will be evaluated for the expression of Hu and other paraneoplastic antigens.
* As part of the study, patients with positive paraneoplastic antibody serology will be requested to undergo a lumbar puncture for antibody determination of these antibodies, cellcount, and chemistry (proteins, glucose, and IgG index) in CSF. In pediatric neuroblastoma patients with stage 4 neuroblastoma the lumbar puncture will be avoided, since there is preliminary evidence suggesting increased risk for leptomeningeal dissemination. Antibody positive patients will be offered quantitative sensory testing for evaluation of subclinical sensory neuronopathy. This test analyzes the minimum increments of sensory stimuli (cold, hot and vibration) required to be noticed by the patient, and compares these results with known normal standard values. The test is given by the clinical neurologist, and does not cause any discomfort.

Conventional nerve conduction studies or EMG are not required, unless the patient has symptoms and signs of neuropathy, or the patient is asymptomatic but the quantitative sensory test is abnormal. In these situations nerve conduction and EMG studies of upper and lower extremities will be obtained. All patients who undergo CSF analysis, will be required to have a blood test (glucose, proteins, and IgG) to be compared with the CSF values and to obtain the IgG index (a measurement of intrathecal synthesis of IgG).

* Patients with positive anti-Mys B antibody serology, or with symptoms suggesting LEMS (proximal weakness, decreased or absent reflexes) will be offered EMG, nerve conduction studies, and repetitive stimulation.
* A random sample of 20% of patients not presenting with positive anti-Hu serology will be offered quantitative sensory testing for evaluation of subclinical sensory neuropathy in order to serve as a control group. Spinal fluid from patients who undergo lumbar puncture for reasons unrelated to anti-Hu serology results (approximately 10-15% of patients) will serve as a control for the spinal fluids obtained from seropositive patients. In these patients a sample of blood will be obtained to measure glucose, proteins, IgG, and IgG index

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous cancers or concurrent cancers. Patient has or may have, newly-diagnosed or recurrent SCLC, or mixed small cell/non small cell lung cancer, or neuroblastoma, or ovarian or breast cancer, or Hodgkin's disease in all cases confirmed by pathological review.

Exclusion Criteria:

* Patient refusal to participate in follow-up clinical evaluations. For minors, parental or guardian refusal.
* Patient refusal to provide blood samples for autoantibody determinations and HLA typing (total 4 tubes).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with previous cancers or concurrent cancers. Patient has or may have, newly-diagnosed or recurrent SCLC, or mixed small cell/non small cell lung cancer, or neuroblastoma, or ovarian or breast cancer, or Hodgkin's disease in all cases confirmed by pathological review.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 1995-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Blood samples for autoantibody determinations and HLA typing and clinical evaluations via Symptom Assessment Scale | 15

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Posner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org